CLINICAL TRIAL: NCT06577324
Title: Effect of a Single Session of Live Group Music Therapy on State Anxiety Levels and Well-being During Chemotherapy: A Multicenter Randomized Clinical Trial
Brief Title: Music Therapy on State Anxiety Levels and Well-being During Chemotherapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Claudia Aristizábal (Other)
Collaborators: SONO (Unknown); keralty (Unknown); Clinica El Carmen (Unknown); Clínica Sebastián de Belalcazar (Unknown)
Responsible Party: Sponsor-Investigator, Claudia Aristizábal, Director, Sanitas University
Organization: Sanitas University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 062-24 UNV
Record Dates: First submitted 2024-08-21; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Anxiety State; Well-Being, Psychological
Keywords: Anxiety; Well-Being; Music Therapy
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Live group music therapy
  Interventions: Behavioral: Live group music therapy
- Non-intervention (No Intervention): Standard health care

INTERVENTIONS:
Behavioral: Live group music therapy — The intervention will involve the use of live music in a group of patients during their quimiotherapy session. The intervention will last approximately forty minutes and will be organized into three stages: Opening (10 min), Body Awareness and Movement (7-10 minutes), Intervention Development (20 minutes). Genres and songs are performed based on the group's preferences and suggestions. The instruments used for the group intervention are the same as those mentioned earlier; participants are provided with percussion instruments, accompanied by the music therapist's voice and the participants' voices. The intervention encourages active participation, with users playing the instruments, singing, engaging in dialogue, and/or reflecting between songs.
  Arms: Intervention

SUMMARY:
Introduction: Many cancer patients experience high levels of anxiety during chemotherapy, which can negatively impact their mental health and physiological, emotional, and spiritual well-being. Various complementary therapies exist to mitigate these effects, including music therapy. Although preliminary evidence supports the positive effects of music therapy and music-based interventions in chemotherapy, few studies report live group interventions conducted by accredited music therapists.

Objective: To determine the effect of a single session of live group music therapy on state anxiety levels and well-being in adult cancer patients undergoing chemotherapy.

Methodology: This study is a multicenter, randomized clinical trial with two arms. The intervention group will receive standard care plus a live group music therapy session, while the control group will receive standard care only. The primary outcome measure is the State-Trait Anxiety Inventory (STAI-E), and the secondary outcome measure is well-being, assessed using the Well-being Numerical Rating Scales (WB-NRSs). The scales will be administered before and after each intervention. The sample size is 102 patients.

Expected Results: This study aims to improve the psycho-emotional health and well-being of cancer patients during chemotherapy, thereby enhancing the quality of care.

DETAILED DESCRIPTION:
Outpatient chemotherapy rooms are spaces where patients diagnosed with cancer receive their treatment. Chemotherapy poses a significant challenge for many patients and is associated with high levels of pain, anxiety, and depression. Several studies have shown that high levels of anxiety influence patients' physical symptoms, such as nausea and vomiting before and after treatment, revealing that 60% of patients undergoing chemotherapy experience these symptoms. These anxiety levels also affect the activation of the sympathetic nervous system, the release of norepinephrine and adrenaline, and an increase in heart rate, respiratory rate, and blood pressure. For many patients, chemotherapy also disrupts social relationships, generates feelings of hopelessness and emotional vulnerability, and causes a rupture and imbalance in all vital dimensions. Additionally, patients with symptoms of depression and anxiety perceive the side effects of chemotherapy more intensely, which significantly impacts their quality of life. This is crucial because it highlights that the patient's mental health and well-being directly influence the course of their illness and their ability to tolerate treatment.

Furthermore, secondary factors such as waiting times both in waiting rooms and within the chemotherapy room can also generate fear, uncertainty, anxiety, discomfort, anger, and irritability. Notably, the environment of the room, filled with different types of noises and sounds, can also affect the mental health of patients.

Due to all of the above, there is a need to explore new strategies to support the chemotherapy process and improve patients' quality of life. Music therapy is one of these strategies, and preliminary evidence suggests it may reduce anxiety symptoms and positively impact the side effects of chemotherapy. Listening to and performing music has a direct effect on the limbic system and can help lower cortisol levels and increase endorphin production.

This research proposal aims to determine the effect of group music therapy on the state anxiety levels and well-being of adult oncology patients attending the chemotherapy rooms at the Sebastián de Belalcázar Clinic in Cali and the El Carmen Clinic in Barranquilla.

Research Question: What is the effect of a single live group music therapy intervention on the state anxiety levels and well-being of adult patients with any type of oncological condition during chemotherapy at the Sebastián de Belalcázar Clinic and the El Carmen Clinic?

ELIGIBILITY:
Inclusion Criteria:

* Patients with a cancer diagnosis, attending intravenous chemotherapy sessions at the Sebastián de Belalcázar and del Carmen clinics.
* Patients over 18 years old.
* Patients who have never previously received music therapy.
* Patients with literacy skills.

Exclusion Criteria:

* Patients who report having hearing problems.
* Patients who express a desire not to participate in the study.
* Patients with difficulties understanding and completing questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
State-trait Anxiety | Baseline and immediately after the intervention
  State-trait Anxiety will be assessed pre and post intervention. To measure state anxiety levels, the STAI (State-Trait Anxiety Inventory) scale will be used. This scale consists of 40 items scored using a Likert scale with four response options (0-3). Twenty items measure trait anxiety (STAI-T) and the other twenty measure state anxiety (STAI-S). Due to the nature of this study, only state anxiety levels will be measured. The Spanish version of the scale has been validated, with a Cronbach's alpha internal consistency ranging from 0.9 to 0.93, and it has demonstrated adequate reliability and validity. The STAI-S will be administered before and after each intervention.

SECONDARY OUTCOMES:
Wellbeing | Baseline and immediately after the intervention
  To measure well-being levels, the WB-NRSs (The Well-Being Numerical Rating Scales) will be used. These scales assess well-being across five different dimensions: physical, psychological, social, spiritual, and general well-being. Each of these domains is measured using a visual analog scale with a score ranging from 1 to 10. The Spanish validation is currently in publication. The WB-NRSs will be administered before and after each intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ettenberg, PhD, Principal Investigator — SONO
Locations (1):
- Clínica Colsanitas, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reyes Aragon L, Diaz AM, Suarez R, Amarillo MA, Colmenares Mejia CC, Ettenberger M. Effect of a Single Live Group Music Therapy Intervention on Anxiety-State and Well-Being Levels During Chemotherapy: A Multicenter Randomized Clinical Trial Protocol. Glob Adv Integr Med Health. 2024 Dec 26;13:27536130241310241. doi: 10.1177/27536130241310241. eCollection 2024 Jan-Dec. PMID 39737328